CLINICAL TRIAL: NCT02171208
Title: A Randomized, Double-Blind, Crossover Study in Healthy Volunteers to Establish the Bioequivalence of BG00012 Supplied by 2 Different Commercial Manufacturers (Vifor SA and Biogen Idec OSD)
Brief Title: A Healthy Volunteer Study to Establish the Bioequivalence of BG00012 Supplied by 2 Different Commercial Manufacturers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 109HV112
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
MeSH Terms: interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference, Test, Reference (RTR) (Active Comparator): Doses will be separated by a washout period
  Interventions: Drug: dimethyl fumarate - Reference form; Drug: dimethyl fumarate - Test form
- Test, Reference, Reference (TRR) (Active Comparator): Doses will be separated by a washout period
  Interventions: Drug: dimethyl fumarate - Reference form; Drug: dimethyl fumarate - Test form

INTERVENTIONS:
Drug: dimethyl fumarate - Reference form — single dose 240 mg
  Other Names: BG00012 Tecfidera®
Drug: dimethyl fumarate - Test form — single dose 240 mg
  Other Names: BG00012

SUMMARY:
The primary objective of this study is to establish the bioequivalence of the test product (BG00012 [dimethyl fumarate] supplied by Biogen Idec OSD) to the reference product (BG00012 supplied by Vifor SA) by comparison of pharmacokinetic (PK) profiles in healthy volunteers.

The secondary objectives of this study are to determine the safety and tolerability of the test product compared to the reference product, to estimate PK parameters of the test product and the reference product, and to estimate the intra-subject coefficient of variation (CV%) of the referenced product for both area under the plasma concentration curve (AUC) and peak plasma concentration (Cmax).

ELIGIBILITY:
Key Inclusion Criteria:

* BMI of 19.0 to 30.0 kg/m2, inclusive
* Subjects of reproductive potential must agree to practice effective contraception from at least 14 days prior to the first dose of study drug through at least 30 days after their last dose of study drug.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, GI, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
* Treatment with another investigational drug or approved therapy for investigational use within 30 days (or 5 half-lives, whichever is longer) prior to Day -1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUCinf) of BG00012 | Up to 48 hours following each dose administration
Maximum observed concentration (Cmax) of BG00012 | Up to 48 hours following each dose administration

SECONDARY OUTCOMES:
The number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 13
Area under the plasma concentration curve from time of dosing to 48 hours | Up to 48 hours following each dose administration
Apparent clearance (CL/F) | Up to 48 hours following each dose administration
Time to peak plasma concentration (Tmax) | Up to 48 hours following each dose administration
Lag time (tlag) | Up to 48 hours following each dose administration
Half-life (t1/2) | Up to 48 hours following each dose administration
Intra-subject coefficient of variation (CV%) of the reference product for area under the plasma concentration curve (AUC) and peak plasma concentration (Cmax) | Up to 48 hours following each dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Research Site, Daytona Beach, Florida
  - Research Site, Evansville, Indiana